CLINICAL TRIAL: NCT00663169
Title: A Randomized, Double-blind, Double-dummy, Active-controlled, Parallel Group Study of a Single Dose of ACZ885 in Hospitalized Patients With Acute Gout
Brief Title: Efficacy and Safety of a Single Dose of Canakinumab (ACZ885) in Hospitalized Patients With Acute Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885A2212
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-12

CONDITIONS: Arthritis, Gouty
Keywords: Arthritis Gouty; ACZ885; IL1B protein; Pain
MeSH Terms: conditions — Arthritis, Gouty; Pain | interventions — canakinumab; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canakinumab (Experimental): Canakinumab 10 mg/kg intravenous infusion and placebo matching dexamethasone intravenous infusion on Day 1.
  Interventions: Biological: canakinumab; Other: placebo matching dexamethasone
- Dexamethasone (Active Comparator): Dexamethasone 12 mg intravenous infusion and placebo matching canakinumab on Day 1.
  Interventions: Drug: dexamethasone; Other: placebo matching canakinumab

INTERVENTIONS:
Biological: canakinumab — 10 mg/kg intravenous infusion 250 mL over 2 hours.
  Other Names: ACZ885; Ilaris®
  Arms: Canakinumab
Drug: dexamethasone — 12 mg intravenous infusion 50 mL over 30 minutes.
  Arms: Dexamethasone
Other: placebo matching canakinumab — 5% glucose in water intravenous infusion.
  Arms: Dexamethasone
Other: placebo matching dexamethasone — Placebo intravenous infusion.
  Arms: Canakinumab

SUMMARY:
This is an exploratory proof-of-concept study to evaluate the safety and efficacy of canakinumab (ACZ885) for inflammation and pain associated with acute gouty arthritis.

ELIGIBILITY:
Inclusion Criteria:

* score over 50 on the 0-100 VAS pain scale
* acute, confirmed gout flare for no longer than 3 days

Exclusion Criteria:

* Treatment with biological anti-tumor necrosis factor (anti-TNF) within the past 3 months
* Anti-inflammatory medication for the treatment of acute gout within the previous 24 hours
* Pregnant or breastfeeding women
* Major surgery with high infection risk
* History of severe allergy to food or drugs
* History or risk of tuberculosis
* Active infection

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (4):
- United States (2):
  - Novartis Investigator Site, Birmingham, Alabama
  - Novartis Investigator Site, New Brunswick, New Jersey
- Novartis Investigator Site, Lausanne, Switzerland
- Novartis Investigator Site, Glasgow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Canakinumab | Dexamethasone
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab | Dexamethasone | Total
Number analyzed (Participants) | 3 | 3 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 46.7 (10.97) | 46.0 (3.46) | 46.3 (7.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Improvement in Gout at 72 Hours Post-dose Using a Likert Scale
Description: 72 hours following treatment, patients were asked the question: "How would you rate the improvement in your gout since receiving the study medication?" Patients rated their improvement on the Likert 5-point scale: 1=Excellent, 2=Good, 3=Acceptable,4=Slight and 5=Poor. Improvement was assessed by determining patients who scored a "good" or "excellent" response.
Time Frame: 72 hours
Population: Pharmacodynamic set included all randomized subjects with evaluable (or complete) pharmacodynamic parameter data.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab | Dexamethasone
Number analyzed (Participants) | 3 | 3
Percentage of participants | 100 | 100

2. Secondary Outcome: Non-inferiority of a Single Dose of Canakinumab Compared to Dexamethasone During Treatment Period
Time Frame: 72 hours
Population: Since the study only recruited 6 subjects this analysis was not done.
Arm/Group | Canakinumab | Dexamethasone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Recurrence of the Symptoms of Acute Gout (if Applicable) During Treatment Period
Description: Time to recurrence is defined as from the point of improvement (good to excellent on Likert scale) to recurrence.
Time Frame: 4 months
Population: Since the study recruited only 6 subjects this analysis was not done.
Arm/Group | Canakinumab | Dexamethasone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Walk Independently (if Applicable) During Treatment Period
Time Frame: 4 months
Population: Since the study recruited only 6 subjects this analysis was not done.
Arm/Group | Canakinumab | Dexamethasone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Discontinuation of Treatment Due to Adverse Events, Deaths or Serious Adverse Events During the Study
Description: Additional safety information can be found in the Adverse Event section.
Time Frame: 4 months
Measure: Number; unit: Participants
Arm/Group | Canakinumab | Dexamethasone
Number analyzed (Participants) | 3 | 3
Participants
  Discontinuation from treatment | 0 | 0
  Death | 0 | 0
  Serious Adverse Event | 0 | 1

6. Secondary Outcome: Change in C-reactive Protein (CRP) From Baseline at Month 4
Description: Blood was collected at Baseline and Month 4 for CRP to identify the presence of inflammation, to determine its severity, and to monitor response to treatment. A negative change from baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: Pharmacodynamic set included all randomized patients with evaluable (or complete) pharmacodynamic parameter data.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Canakinumab | Dexamethasone
Number analyzed (Participants) | 3 | 3
mg/L | -22.23 (16.822) | -30.30 (51.963)

7. Secondary Outcome: Change in Serum Amyloid A Protein (SAA) From Baseline at Month 4
Description: Blood was collected at Baseline and Month 4 for SAA to identify the presence of inflammation, to determine its severity, and to monitor response to treatment. A negative change from baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: Pharmacodynamic set included all randomized patients with evaluable (or complete) pharmacodynamic parameter data.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Canakinumab | Dexamethasone
Number analyzed (Participants) | 3 | 3
mg/L | -579.980 (563.7449) | -260.327 (463.8600)

8. Secondary Outcome: ACZ885 (Canakinumab) Pharmacokinetics (PK) Serum Concentration During the Treatment Period
Description: Blood was collected for ACZ885 (canakinumab) levels at baseline and Days 0.25, 1, 3, 6, 20, 34, 55 and 119. Serum was analyzed by means of a competitive Enzyme linked immunosorbant assay (ELISA).
Time Frame: Baseline, Days 0.25, 1, 3, 6, 20, 34, 55 and 119
Population: Pharmacodynamic set included all randomized subjects with evaluable (or complete) pharmacodynamic parameter data.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Canakinumab
Number analyzed (Participants) | 3
μg/mL
  Baseline | 0.0 (0.00)
  Day 0.25 | 221.5 (143.58)
  Day 1 (n=2) | 276.5 (26.163)
  Day 3 (n=1) | 92.3 (NA) — Standard deviation not calculated- data available for only 1 participant.
  Day 6 | 136.6 (41,532)
  Day 20 | 72.37 (11.154)
  Day 34 | 52.87 (13.194)
  Day 55 | 31.67 (8.4884)
  Day 119 | 7.643 (4.6151)

9. Secondary Outcome: Change From Baseline in Pain Using a Visual Analog Scale at Month 4
Description: Patients rated their pain on a 100 millimeter (mm) visual analog scale, ranging from no pain (0) to unbearable pain (100). A negative change from baseline indicates improvement.
Time Frame: Baseline, Month 4
Population: Pharmacodynamic set included all randomized subjects with evaluable (or complete) pharmacodynamic parameter data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Canakinumab | Dexamethasone
Number analyzed (Participants) | 3 | 3
Score on a scale | -62.0 (3.61) | -65.7 (17.62)

10. Secondary Outcome: Number of Patients Who Took Rescue Medication
Description: Patients who did not improve by 72 hours post-dose (i.e. patients who show a pain Visual Analog (VAS) decrease of less than 50 % from baseline (Day 1, pre-dose) would have been treated with rescue medication of methylprednisolone 80 mg intravenous or intramuscular once at the discretion of the clinical investigator.
Time Frame: 4 months
Population: All participants.
Measure: Number; unit: Participants
Arm/Group | Canakinumab | Dexamethasone
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Canakinumab | Dexamethasone
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=3) | Dexamethasone (N=3)
Gout (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=3) | Dexamethasone (N=3)
Ocular hyperaemia (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.